CLINICAL TRIAL: NCT03461445
Title: A Pilot Study to Evaluate Impact on Neurological Side Effects (Cognition, Memory, and Tremor) in Elderly (Age>65) Patients
Brief Title: Effect of Tacrolimus Formulation on Neurological Side Effects in Older Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1044220
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplant; Complications; Toxicity; Drug Toxicity; Neurotoxicity
Keywords: Elderly; Neurotoxicity; Calcineurin inhibitors; Tacrolimus
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Neurotoxicity Syndromes | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Release Tacrolimus (Active Comparator): Patients will receive immediate release tacrolimus
  Interventions: Drug: IR Tacrolimus
- Envarsus (Experimental): Patients will be converted to Envarsus formulation of tacrolimus
  Interventions: Drug: Envarsus

INTERVENTIONS:
Drug: Envarsus — Patients will be randomized to receiving Envarsus instead of IR Tacrolimus
  Arms: Envarsus
Drug: IR Tacrolimus — Patients will be randomized to receiving IR Tacrolimus instead of Envarsus
  Arms: Immediate Release Tacrolimus

SUMMARY:
Previous studies have shown that elderly patients experience higher trough levels of tacrolimus and are more sensitive to the effects of medications, they experience higher occurrence and severity of such medication related toxicities. Therefore, the investigators hypothesize that by transitioning patients from tacrolimus immediate release to Envarsus ®, the peak-dose effect will be eliminated or attenuated, leading to a significant decrease in neurocognitive toxicities in the older patient population.

DETAILED DESCRIPTION:
The investigators will conduct a single-center, prospective, open-label, randomized study to evaluate the difference in neurocognitive side effects between Envarsus and immediate release tacrolimus. Eligible patients will be enrolled within 8 weeks post-transplantation. They will be administered a baseline panel of neurocognitive tests. They will then be randomized to either continue on immediate release tacrolimus or Envarsus. 6 weeks after randomization, the neurocognitive tests will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of a kidney transplant
2. Age 60 or greater at the time of transplant
3. Kidney graft is functional (not dialysis dependent) by 4 weeks post-transplant
4. Have IR tacrolimus as maintenance therapy
5. Have BMI < 35 at time of transplant
6. Achieve therapeutic tacrolimus level within 4 weeks post-transplant

Exclusion Criteria:

1. Recipient of a simultaneous non-kidney transplant (pancreas)
2. Had an episode of rejection before study enrollment
3. Had a TIA/CVA after transplantation and before study enrollment
4. Had a neurologic injury after transplantation and before study enrollment
5. Blindness
6. Have an mTOR inhibitor as maintenance therapy
7. Nonadherence, as determined by a trough level less than 7 ng/mL after achieving therapeutic level with no other rationale for sub-therapeutic levels.
8. Adults unable to consent
9. Pregnant women
10. Prisoners

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Xin Chen, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/an-experimental-comparison-study-of-envarsus-xr-and-tacrolimus-ir-for-elderly-kidney-transplant-patients-443391/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Release Tacrolimus | Envarsus
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Release Tacrolimus | Envarsus | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (5.4) | 69 (4.2) | 69 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 10 | 25
  Black | 0 | 3 | 3
  Asian | 4 | 6 | 10
  Hispanic | 12 | 7 | 19
  Multi-racial | 0 | 1 | 1
  Unknown/Other | 1 | 2 | 3
  Native Hawaiian / Pacific Islander | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurocognitive Side Effects
Description: Change in MOCA (Montreal Cognitive Assessment) from baseline to study end. MOCA scale runs from 0 to 30 with higher being a better outcome.
  Change in DSST (Digital Symbol Substitution Test) from baseline to study end. DSST scale runs from 1 to 125 with higher being a better outcome.
Time Frame: 6 weeks after randomization and baseline testing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Release Tacrolimus | Envarsus
Number analyzed (Participants) | 31 | 31
score on a scale
  MOCA score difference | 1.2 (2.1) | 0.2 (2.9)
  DSST score difference | 1.0 (7.8) | 1.26 (7.5)

2. Secondary Outcome: Change in Self-reported Side Effects
Description: Quality of life in Essential Tremor questionnaire (QUEST) Summary Score: A 30-item scale assessing the impact of tremor on various domains of quality of life, such as communication, work and hobbies. In the QUEST questionnaire scale, a lower score is indicative of better quality of life while higher scores indicate poorer quality of life. The score is a percentage ranging from zero to 100.
Time Frame: 6 weeks after randomization and baseline testing
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Immediate Release Tacrolimus: Individuals taking immediate release tacrolimus
- LCP Tacrolimus: Individuals taking prolonged release tacrolimus
Arm/Group | Immediate Release Tacrolimus | LCP Tacrolimus
Number analyzed (Participants) | 32 | 32
score on a scale | -1.2 (7.5) | -3.1 (9)

3. Secondary Outcome: Kidney Graft Survival
Description: Number of kidney grafts still functioning at the end of the study
Time Frame: 6 months after transplant
Measure: Number; unit: kidney grafts
Arm/Group | Immediate Release Tacrolimus | LCP Tacrolimus
Number analyzed (Participants) | 32 | 32
kidney grafts | 32 | 32

4. Secondary Outcome: Patient Survival
Description: Number patients who survived during the study
Time Frame: 6 months after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Release Tacrolimus | LCP Tacrolimus
Number analyzed (Participants) | 32 | 32
Participants | 32 | 32

ADVERSE EVENTS:
Time Frame: While participants were enrolled in the study (6 week period for each individual).
Arm/Group | Immediate Release Tacrolimus | Envarsus
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 2/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Release Tacrolimus (N=32) | Envarsus (N=32)
Cognitive decline (Nervous system disorders) | 0 (0) | 1 (1)
Medication Overdose (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03461445/Prot_SAP_002.pdf